CLINICAL TRIAL: NCT05269186
Title: Interest of Virtual Reality on Anxiety Before the Planning CT Scan in Radiotherapy
Acronym: REAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHD22_0002
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Pelvic Cancer
MeSH Terms: conditions — Breast Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Virtual reality session performed before the planning CT scan
  Interventions: Device: Virtual reality software
- Normal care (No Intervention): Normal care without intervention

INTERVENTIONS:
Device: Virtual reality software — The patient will undergo a 20-minute virtual reality session before the planning CT scan
  Arms: Virtual reality

SUMMARY:
In France, according to the National Cancer Institute, it appears that treatments in radiotherapy centers for cancer will increase from 198,000 in 2015 to 239,000 in 2030: this represents 40,000 additional treatments in 15 years.

A meta-analysis on radiotherapy indicated that 10 to 20% of patients had clinically significant levels of anxiety at the beginning of radiotherapy.

Indeed, several factors generate this tension, above all the new or unfamiliar environment, the imposing and noisy scanner, the restraints that are difficult to bear or the nudity required for the examination.

This anxiety has an impact on performance of the planning CT scan examination, an essential step for the future treatment.

The radiotherapy unit of the Centre Hospitalier Departemental de Vendee has put in place resources to reduce anxiety felt during treatment sessions (music therapy, conversational hypnosis, sophrology or aromatherapy). However, nothing has been put in place to reduce the anxiety of patients in the period preceding the planning CT scan.

Virtual reality software seems to be a good alternative that requires fewer human resources.

The research hypothesis is that patients who have benefited from the virtual reality software will have a lower level of anxiety before the planning CT scan than patients who have not benefited from virtual reality.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an indication for first radiotherapy treatment for breast or pelvic cancer (prostate, rectum, endometrium, anal canal and cervix)
2. Patient ≥ 18 years old,
3. Patient who has the capacity to understand the protocol and has given written consent to participate in the research,
4. Patient with social security coverage.

Exclusion Criteria:

1. Metastatic patients
2. Patients with previous radiotherapy
3. Patients with a diagnosis of hearing impairment
4. Patients with major cognitive disorders (such as dementia)
5. Psychiatric pathology such as schizophrenia
6. Patients with epilepsy or hypersensitivity to flashing lights
7. Patient with a pacemaker, hearing aid or defibrillator
8. Claustrophobic patients
9. Patients sensitive to motion sickness
10. Patients who are visually impaired or blind
11. Patients with migraine
12. Patients with skin defects and open wounds in the area where the helmet is applied (face or scalp) or in the eyes
13. Patients under guardianship, curators or deprived of liberty
14. Non French speaking patient
15. Illiterate patient
16. Patient participating in another clinical investigation or interventional clinical research protocol involving a drug
17. Pregnant or breastfeeding patient

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Evaluating the anxiety of the patient benefiting from a virtual reality session versus normal care management | 10 minute before the planning CT scan
  Anxiety level measured by the State Anxiety Scale of Spielberger. The scale is a validated 20 item self report assessment device. The score range is 20-80, the higher score indicating anxiety. The cut point of 39-40 has been suggested to detect clinically significant symptoms for the State Anxiety scale.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa ZINZONI, Principal Investigator — vanessa.zinzoni@ght85.fr
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No